CLINICAL TRIAL: NCT03317197
Title: Comparison of the Effect of Vasopressin, Steroid, and Epinephrine Treatment in Patients With Out-of-hospital Cardiac Arrest: Multi-center, Double Blind, Randomized, Placebo-controlled Study
Brief Title: Effect of Vasopressin, Steroid, and Epinephrine Treatment in Patients With Out-of-hospital Cardiac Arrest
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Jung-Youn Kim, Assistant Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: KUGH17156 (VSE study)
Record Dates: First submitted 2017-10-04; First posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Cardiac Arrest
Keywords: Out-of-Hospital Cardiac Arrest; Vasopressin-steroid-epinephrine (VSE); Treatment Outcome; prognosis; Return of spontaneous circulation
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest | interventions — Control Groups; Epinephrine; Vasopressins; Steroids

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (Placebo Comparator): * Using Epinephrine(1 mg/cardiopulmonary resuscitation(CPR) cycle) only
  * Control group receives intravenous injection of 1 mg epinephrine every cycle (about 3 minutes) during CPR and uses syringe No. 1, 5 times (every 3 minutes), and syringe No. 2, one time (in the first cycle). After each injection, inject 10 mL saline solution additionally.
    * Syringe No. 1 : Saline solution
    * Syringe No. 2 : Saline solution
  Interventions: Drug: Control Group
- Experimental Group 1 (Active Comparator): * Using Vasopressin [20 IU/CPR cycle] injection until the 5th cycle
  * Experimental Group 1 receives intravenous injection of 1 mg epinephrine every cycle (about 3 minutes) during CPR and uses syringe No. 1, 5 times (every 3 minutes), and syringe No. 2, one time (in the first cycle). After each injection, inject 10 mL saline solution additionally.
    * Syringe No. 1 : Vasopressin
    * Syringe No. 2 : Saline solution
  Interventions: Drug: Experimental Group 1
- Experimental Group 2 (Active Comparator): * Using Epinephrine(1 mg/cardiopulmonary resuscitation(CPR) cycle) and Steroid(Methylprednisolone, 40 mg at first cycle)
  * Experimental Group 2 receives intravenous injection of 1 mg epinephrine every cycle (about 3 minutes) during CPR and uses syringe No. 1, 5 times (every 3 minutes), and syringe No. 2, one time (in the first cycle). After each injection, inject 10 mL saline solution additionally.
    * Syringe No. 1 : Saline solution
    * Syringe No. 2 : Steroid
  Interventions: Drug: Experimental Group 2
- Experimental Group 3 (Experimental): * Using Epinephrine(1 mg/cardiopulmonary resuscitation(CPR) cycle), Vasopressin(20 international unit(IU)/cardiopulmonary resuscitation(CPR) cycle) and Steroid(Methylprednisolone, 40 mg at first cycle)
  * Experimental Group 3 receives intravenous injection of 1 mg epinephrine every cycle (about 3 minutes) during CPR and uses syringe No. 1, 5 times (every 3 minutes), and syringe No. 2, one time (in the first cycle). After each injection, inject 10 mL saline solution additionally.
    * Syringe No. 1 : Vasopressin
    * Syringe No. 2 : Steroid
  Interventions: Drug: Experimental Group 3

INTERVENTIONS:
Drug: Control Group — Using Epinephrine(1 mg/cardiopulmonary resuscitation(CPR) cycle) only
  Other Names: Epinephrine
  Arms: Control Group
Drug: Experimental Group 1 — Using Epinephrine(1 mg/cardiopulmonary resuscitation(CPR) cycle) and Vasopressin(20 international unit(IU)/cardiopulmonary resuscitation(CPR) cycle)
  Other Names: Epinephrine + Vasopressin
  Arms: Experimental Group 1
Drug: Experimental Group 2 — Using Epinephrine(1 mg/cardiopulmonary resuscitation(CPR) cycle) and Steroid(Methylprednisolone, 40 mg at first cycle)
  Other Names: Epinephrine + Steroid
  Arms: Experimental Group 2
Drug: Experimental Group 3 — Using Epinephrine(1 mg/cardiopulmonary resuscitation(CPR) cycle), Vasopressin(20 international unit(IU)/cardiopulmonary resuscitation(CPR) cycle) and Steroid(Methylprednisolone, 40 mg at first cycle)
  Other Names: Epinephrine + Vasopressin + Steroid
  Arms: Experimental Group 3

SUMMARY:
Steroid use could be considered for patients with weaker adrenal function among those with post-cardiac arrest (CA) return of spontaneous circulation (ROSC), according to the former study. This finding is consistent with the medical background of this present study. This study will be the first to investigate these additional drugs of injection and associated prognosis in cardiac arrest (CA) patients outside the hospital, providing significant basic data.

DETAILED DESCRIPTION:
In South Korea, approximately 20,000 patients are found to experience cardiac arrest (CA) annually, with a reported survival rate of approximately 4.8% (2015). In patients who are resuscitated from cardiac arrest (CA), neurological prognosis is assessed based on whether the patient can independently perform a daily routine after leaving the hospital. It is an essential issue for patients, as well as their families and local communities. In this sense, research interest in achieving a good neurological prognosis in post-discharge cardiac arrest (CA) patients is increasing. The neurologic status of post-cardiac arrest (CA) patients, who are being considered for discharge from the hospital, is examined mostly using the Cerebral Performance Category (CPC) score, with a score of 1 or 2, on a scale of 1 to 5, indicative of good neurological status.

Several previous South Korean studies have compared treatments using epinephrine only with those using epinephrine, vasopressin, and steroid during cardiopulmonary resuscitation (CPR) of cardiac arrest (CA)patients in the hospital. The vasopressin-steroid-epinephrine (VSE) group was reported to show a better return of spontaneous circulation (ROSC), lower whole-body inflammatory reaction, less cases of organ failure, and more cases of survival and hospital leave while showing better results of neurological prognosis. However, studies are lacking on treatment of cardiac arrest (CA) cases outside the hospital. In addition, because the three drugs of the vasopressin-steroid-epinephrine (VSE) regimen are used together, it is hard to identify which of them is most effective. Investigators are implementing a multicenter, prospective study to compare the use of vasopressin, steroid, and both vasopressin and steroid in post-cardiac arrest (CA) patients outside the hospital and examine the effects on ROSC and neurological score in this population.

No South Korean study has been conducted on additional drugs of injection, other than epinephrine, in cardiac arrest (CA) treatment. In one study, steroid use in post-cardiac arrest (CA) patients with return of spontaneous circulation (ROSC) was investigated by examining the levels of blood cortisol and adrenal corticotropic hormone. The researchers found that patients showing relatively poorer results in the exams recorded lower. Therefore, steroid use could be considered for patients with weaker adrenal function among those with post-cardiac arrest (CA) return of spontaneous circulation (ROSC), according to the study.

This finding is consistent with the medical background of this present study. It is possible that steroid use not only assists the adrenal function in post-cardiac arrest (CA) patients but also positively influences their spontaneous circulation recovery and neurological prognosis. However, this research is also the result of a single-organizational retrospective study. To establish additional corresponding experiences, a multicenter prospective investigation is deemed necessary.

As previously mentioned, several studies involving in-hospital cardiac arrest (CA) patients have been conducted. The present study will be the first to investigate these additional drugs of injection and associated prognosis in cardiac arrest (CA) patients outside the hospital, providing significant basic data.

ELIGIBILITY:
Inclusion Criteria:

* The group of patients who participated in the study included adults aged at least 19 years among the atraumatic CA outpatients who came to the ER and received CPR.

Exclusion Criteria:

* Pregnant women and young children aged <18 years;
* Patients with underlying disease cases without the possibility of resuscitation (e.g., terminal cancer);
* Patients with do-not-resuscitate (DNR) status;
* Death by excessive bleeding (e.g., abdominal main artery rupture);
* Patients who have experienced in-hospital CA;
* Patients previously treated with steroid, anti-cancer medicine, or immunosuppression treatment before CA;
* Patients already been registered with other studies; or
* Patients from whom informed consent cannot be obtained

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 834 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2020-08-09 (Estimated); Study Completion 2020-08-09 (Estimated)

PRIMARY OUTCOMES:
Examined for neurological prognosis of each group | survival discharge, through study completion, an average of 1 year
  - main result variables: survival discharge with good CPC (CPC 1 or 2)

SECONDARY OUTCOMES:
Examined for return of spontaneous circulation (ROSC) status | ROSC, up to 24 hours
  sustained ROSC (more than 20mins)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Youn Kim, MD, Ph.D., Principal Investigator — Assistant Professor
Locations (1):
- Korea University Guro Hospital, Seoul, Guro-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mentzelopoulos SD, Zakynthinos SG, Tzoufi M, Katsios N, Papastylianou A, Gkisioti S, Stathopoulos A, Kollintza A, Stamataki E, Roussos C. Vasopressin, epinephrine, and corticosteroids for in-hospital cardiac arrest. Arch Intern Med. 2009 Jan 12;169(1):15-24. doi: 10.1001/archinternmed.2008.509. PMID 19139319
- [Background] Nolan JP, Deakin CD, Soar J, Bottiger BW, Smith G; European Resuscitation Council. European Resuscitation Council guidelines for resuscitation 2005. Section 4. Adult advanced life support. Resuscitation. 2005 Dec;67 Suppl 1:S39-86. doi: 10.1016/j.resuscitation.2005.10.009. No abstract available. PMID 16321716
- [Background] Mentzelopoulos SD, Malachias S, Chamos C, Konstantopoulos D, Ntaidou T, Papastylianou A, Kolliantzaki I, Theodoridi M, Ischaki H, Makris D, Zakynthinos E, Zintzaras E, Sourlas S, Aloizos S, Zakynthinos SG. Vasopressin, steroids, and epinephrine and neurologically favorable survival after in-hospital cardiac arrest: a randomized clinical trial. JAMA. 2013 Jul 17;310(3):270-9. doi: 10.1001/jama.2013.7832. PMID 23860985
- [Background] Mentzelopoulos SD, Mongardon N, Xanthos T, Zakynthinos SG. Possible significance of hemodynamic and immunomodulatory effects of early stress-dose steroids in cardiac arrest. Crit Care. 2016 Jul 20;20(1):211. doi: 10.1186/s13054-016-1384-4. No abstract available. PMID 27436285
- [Background] Donnino MW, Andersen LW, Berg KM, Chase M, Sherwin R, Smithline H, Carney E, Ngo L, Patel PV, Liu X, Cutlip D, Zimetbaum P, Cocchi MN; Collaborating Authors from the Beth Israel Deaconess Medical Center's Center for Resuscitation Science Research Group. Corticosteroid therapy in refractory shock following cardiac arrest: a randomized, double-blind, placebo-controlled, trial. Crit Care. 2016 Apr 3;20:82. doi: 10.1186/s13054-016-1257-x. PMID 27038920
- [Background] Link MS, Berkow LC, Kudenchuk PJ, Halperin HR, Hess EP, Moitra VK, Neumar RW, O'Neil BJ, Paxton JH, Silvers SM, White RD, Yannopoulos D, Donnino MW. Part 7: Adult Advanced Cardiovascular Life Support: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S444-64. doi: 10.1161/CIR.0000000000000261. No abstract available. PMID 26472995
- [Background] Kim JJ, Lim YS, Shin JH, Yang HJ, Kim JK, Hyun SY, Rhoo I, Hwang SY, Lee G. Relative adrenal insufficiency after cardiac arrest: impact on postresuscitation disease outcome. Am J Emerg Med. 2006 Oct;24(6):684-8. doi: 10.1016/j.ajem.2006.02.017. PMID 16984836
- [Background] Kim JY, Shin SD, Ro YS, Song KJ, Lee EJ, Park CB, Hwang SS; CardioVascular Disease Surveillance (CAVAS) investigators. Post-resuscitation care and outcomes of out-of-hospital cardiac arrest: a nationwide propensity score-matching analysis. Resuscitation. 2013 Aug;84(8):1068-77. doi: 10.1016/j.resuscitation.2013.02.010. Epub 2013 Feb 27. PMID 23454438